CLINICAL TRIAL: NCT03390426
Title: Femoral Peri-arterial Local Anesthetic Injection Decreases Tourniquet Associated Ischemic Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00089161
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Tourniquet Hypertension; Intraoperative Hypertension; Total Ankle Arthroplasty; Ankle Fusion
Keywords: Perifemoral; Tourniquet; Mepivacaine; Tourniquet Hypertension
MeSH Terms: interventions — Mepivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mepivacaine Block Group (Experimental): Injection of local anesthetic (mepivacaine) above and beside the femoral artery.
  Interventions: Drug: Mepivacaine; Procedure: Perifemoral Injection of Local Anesthetic
- Saline Sham Group (Placebo Comparator): Injection of salt water (saline) above and beside the femoral artery.
  Interventions: Procedure: Perifemoral Injection of Local Anesthetic; Drug: Saline

INTERVENTIONS:
Drug: Mepivacaine — An ultrasound guided injection of mepivacaine superomedially to the femoral artery.
  Other Names: Carbocaine
  Arms: Mepivacaine Block Group
Procedure: Perifemoral Injection of Local Anesthetic — An ultrasound guided injection of mepivacaine superomedially to the formal artery in an effort to numb the nerves that contribute to tourniquet hypertension intraoperatively.
  Other Names: Femoral periarterial injection
Drug: Saline — An ultrasound guided injection using a medication that does NOT numb any nerves called saline, or salt water.
  Other Names: Salt Water placebo
  Arms: Saline Sham Group

SUMMARY:
The purpose of this prospective randomized double-blind study is to determine if the novel technique of ultrasound guided peri-arterial injection of local anesthetic around the femoral artery decreases ischemic hypertension associated with prolonged lower extremity tourniquet time during total ankle arthroplasty (TAA) and foot fusion surgeries. Patients will be randomized 1:1 to receive either local anesthetic or saline, which will be injected superomedially to the femoral artery in an attempt to block sympathetic afferents and decrease tourniquet associated hypertension intraoperatively.

DETAILED DESCRIPTION:
The purpose of this prospective randomized double-blind study is to determine if the novel technique of ultrasound guided peri-arterial injection of local anesthetic around the femoral artery decreases ischemic hypertension associated with prolonged lower extremity tourniquet time during total ankle arthroplasty (TAA) and foot fusion surgeries. Efficacy will be determined by analyzing incidence of intraoperative ischemic hypertension, defined as >30% increase in systolic blood pressure, associated with tourniquet inflation times greater than 90 minutes. The study will involve a total of 30 patients (15 in each group) and with a power of 80% to detect a 50% difference. The patients involved in the study will be ASA 1-3 patients who are undergoing either TAA or foot fusion surgeries. Patients will receive standard of care for their anesthesia, which at Duke Hospital includes placement of popliteal and saphenous perineural catheters and a general anesthetic with a laryngeal mask airway. Patients will be randomized to receive femoral peri-arterial injection with either 1.5% mepivacaine with 1:400,000 epinephrine or 0.9% saline which will be performed preoperatively at time of perineural catheter placement. Patients will assume standard risk associated with nerve blocks, including theoretical risk of nerve damage and local anesthetic systemic toxicity. Possible benefits include improved intraoperative hemodynamic stability, decreased intraoperative opioid and antihypertensive medications, and decreased tourniquet associated pain post-operatively.

ELIGIBILITY:
Inclusion Criteria:

Patients that will be included in the study are English speaking 18-75 year old ASA 1-3 patients undergoing total ankle arthroplasty.

Exclusion Criteria:

1. ASA 4 or 5
2. Diagnosis of chronic pain
3. Daily chronic opioid use (over 3 months of continuous opioid use).
4. Inability to communicate pain scores or need for analgesia.
5. Infection at the site of block placement
6. Age under 18 years old or greater than 75 years old
7. Pregnant women (as determined by standard of care day-of surgery urine bHCG)
8. Intolerance/allergy to local anesthetics
9. Weight <50 kg
10. Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
11. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance.
12. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Bullock, Principal Investigator — Assistant Professor
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; patients will be deidentified and no personal information or medical records used.

REFERENCES:
- [Derived] Wahal C, Grant SA, Gadsden J, Rambhia MT, Bullock WM. Femoral artery block (FAB) attenuates thigh tourniquet-induced hypertension: a prospective randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Mar;46(3):228-232. doi: 10.1136/rapm-2020-102113. Epub 2021 Jan 11. PMID 33431616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepivacaine Block Group | Saline Sham Group
Started | 15 | 16
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepivacaine Block Group | Saline Sham Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.47 (11.84) | 65.67 (4.61) | 63.81 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
ASA Status [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) Physical Status Classification. ASA 1 = a normal healthy patient, ASA 2 = a patient with mild systemic disease, ASA 3 = a patient with severe systemic disease.
  Participants
    ASA 1 | 2 | 0 | 2
    ASA 2 | 6 | 7 | 13
    ASA 3 | 7 | 8 | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.11 (4.63) | 32.64 (5.41) | 31.63 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Tourniquet Hypertension
Description: Measuring systolic blood pressure using a cuff, aim to keep <30mmHg change from baseline
Time Frame: Intraoperatively (~3 hours)
Population: Subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepivacaine Block Group | Saline Sham Group
Number analyzed (Participants) | 15 | 15
Participants | 5 | 14

2. Secondary Outcome: Pain Scores as Measured by the Numeric Rating Scale (NRS-11)
Description: The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. 0 = No Pain, 1-3 = Mild Pain, 4-6 = Moderate Pain, 7-10 = Severe Pain.
Time Frame: While in PACU (~1 hour)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mepivacaine Block Group | Saline Sham Group
Number analyzed (Participants) | 15 | 15
score on a scale | 1.80 (2.86) | 1.07 (1.71)

3. Secondary Outcome: Amount of Opioid Pain Medications Used by Patient
Description: Amount of opioid pain medication used by patient over a 4 hour period immediately after surgery. Opioids taken are converted to morphine equivalents.
Time Frame: Perioperative period (~4 hours)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Mepivacaine Block Group | Saline Sham Group
Number analyzed (Participants) | 15 | 15
morphine equivalents | 10.48 (5.77) | 8.19 (4.65)

4. Secondary Outcome: Amount of Esmolol Used Intraoperatively
Description: Amount of esmolol (in mg) used intraoperatively to decrease blood pressure after subject achieved tourniquet hypertension.
Time Frame: Intraoperatively (~3 hours)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Mepivacaine Block Group | Saline Sham Group
Number analyzed (Participants) | 15 | 15
mg | 8.00 (14.24) | 95.33 (107.63)
Statistical Analysis 1: Comparison: Mepivacaine Block Group vs Saline Sham Group; We determined 30 subjects were needed to detect a 50% difference in THN incidence between the two groups using a one-sided Fisher's exact test with alpha = 0.05 and 80% power while allowing up to 20% drop-out. For primary and secondary outcomes, comparisons were made between the two groups using a two-sample t-test or Mann-Whitney U test for continuous variables and Fisher's exact test for categorical variables. p-value of <0.05 was considered to be statistically significant; Test type: Superiority — this is a superiority study and the "non-inferiority or equivalence analysis" is not required; p < 0.05, t-test, 2 sided — Comparisons were made between the two groups using a two-sample t-test or Mann-Whitney U test for continuous variables and Fisher's exact test for categorical variables. p-value of <0.05 was considered to be statistically significant; Comparisons were made using a two-sample t-test or Mann-Whitney U test for continuous variables and Fisher's exact test for categorical variables

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Mepivacaine Block Group | Saline Sham Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03390426/Prot_SAP_000.pdf